CLINICAL TRIAL: NCT02222805
Title: Effect of Timing of Umbilical Cord Clamping on Anaemia at 8 and 12 Months and Later Neurodevelopment in Late Pre-term and Term Infants; a Facility-based Randomized-controlled Trial in Nepal
Brief Title: Effect of Timing of Umbilical Cord Clamping on Anaemia at 8 and 12 Months and Later Neurodevelopment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: UNICEF (Other); Ministry of Health and Population, Nepal (Other Government); The Swedish Society of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CCANEMIA11
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Anemia; Iron Deficiency; Neonatal Jaundice
Keywords: Cord clamping; Iron deficiency; Anemia; Iron; Hyperbilirubinemia; Jaundice; Neurodevelopment
MeSH Terms: conditions — Anemia; Iron Deficiencies; Jaundice, Neonatal; Hyperbilirubinemia; Jaundice | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early cord clamping (ECC) (Other): Early (≤30 seconds) cord clamping of the umbilical cord after delivery.
  Interventions: Procedure: Early (≤30 seconds) cord clamping
- Delayed cord clamping (DCC) (Other): Delayed (≤180 seconds) cord clamping of the umbilical cord after delivery.
  Interventions: Procedure: Delayed (≤180 seconds) cord clamping

INTERVENTIONS:
Procedure: Early (≤30 seconds) cord clamping — Early (≤30 seconds) cord clamping of the umbilical cord after delivery.
  Other Names: Immediate cord clamping
  Arms: Early cord clamping (ECC)
Procedure: Delayed (≤180 seconds) cord clamping — Delayed (≤180 seconds) cord clamping of the umbilical cord after delivery.
  Other Names: Late cord clamping; Deferred cord clamping; Optimal cord clamping
  Arms: Delayed cord clamping (DCC)

SUMMARY:
The investigators plan a study to randomize 540 children in Nepal to early (≤30 seconds) or late (≥180 seconds) clamping of the umbilical cord at birth. The children will be followed with blood tests (hemoglobin and ferritin) at 8 and 12 months of age, and their development is evaluated by questionnaire (Ages & Stages Questionnaire ) at 12 months of age, and by testing (Bayley -III) at 18-24 months of age. By implementing the project in a country with a high proportion of anemia at one year of age (about 75%), we can reduce the number of children in the study and still achieve significant results.

Iron deficiency is a global health problem and causes anemia and impaired neurodevelopment in children. Anemia is estimated by WHO to occur among 25% of all children before school age, and the corresponding figure in Europe is 3-9 %.

By waiting 3 minutes to clamp the cord after birth, a large part of the child's blood volume remaining in the placenta is transfused over to the child's body. Research shows that the neonate's blood volume can increase by about 40% and this blood contains 3 to 4 months' supply of iron. In Sweden, we have shown that late clamping of the umbilical cord could reduce iron deficiency in children at four months of age by 90%. Globally, most countries practice early cord clamping and the child is deprived of the placental blood transfusion. The hypothesis of the study is that by delaying the clamping of the umbilical cord, anemia at 8 and 12 months will be reduced an this in turn will be beneficial for the childrens development.

The project will be implemented at Paropakar Maternity and Women 's Hospital, Kathmandu. It hosts approximately 23,000 births annually.

DETAILED DESCRIPTION:
Study Protocol Effect of timing of umbilical cord clamping on anaemia at 8 and 12 months and later neurodevelopment in late pre-term and term infants; a facility-based randomized-controlled trial in Nepal

Introduction At the time of birth, the infant is still attached to the placenta via the umbilical cord. The infant is usually separated from the placenta by clamping the cord with two clamps. This task takes place during the third stage of labour, which is the period of time from the birth of the infant to the delivery of the placenta.

Active management of the third stage of labour has been described in a recent World Health Organization (WHO) report as the "cornerstone" of obstetric and midwifery practice during the latter part of the 20th century. Active management has involved the clinician intervening in the process through three interrelated processes: the administration of an uterotonic drug; early cord clamping and cutting; and controlled traction of the umbilical cord.

Early cord clamping has been generally advised to be carried out in the first 30 seconds after birth, regardless of whether the cord pulsation has ceased. Due to evidence shown the last decade, recent guidelines for management of the third stage of labour no longer recommend immediate cord clamping but changes in practice is questioned and policies on hospitals are rare.

Possible beneficial and adverse effects:

Delayed clamping allows time for a transfer of the fetal blood in the placenta to the infant at the time of birth. This placental transfusion can provide the infant with an additional 40% more blood volume. The amount of blood returned to the infant depends on when the cord is clamped and at what level the infant is held prior to clamping. Neonatal benefits associated with this increased placental transfusion include higher haemoglobin concentrations, additional iron stores and less anaemia later in infancy, higher red blood cell flow to vital organs and better cardiopulmonary adaptation.

Delayed cord clamping has been linked to an increase in the incidence of jaundice which, in severe cases, could have longer term effects on the health and development of the infant.

Previous studies performed by the principal investigator in a high-income country has shown that delayed cord clamping, compared with early clamping, resulted in reduced prevalence of neonatal anaemia. Furthermore delayed, cord clamping improved iron status and reduced prevalence of iron deficiency (ID) at 4 months of age without demonstrable adverse effects. As ID in infants even without anaemia has been associated with impaired development , delayed cord clamping seems to benefit full term infants even in regions with a relatively low prevalence of ID anaemia.

Later effects on anaemia and development:

The improved iron stores at four to six months after delayed cord clamping suggests that ID anaemia could be reduced at eight to twelve months of age, but this could not be shown in the principal investigators latest study, possibly due to small sample size. Although ID anaemia is rare (3-9 %) in high income countries, the negative impact on children's health and development should not be underestimated. As an example, a 15 % reduction of anaemia in Sweden among toddlers (from 3 to 2,5 %) would help 500 children annually. No randomized trial has evaluated the effect of delayed versus early cord clamping on infants after 6 months of age in a low income country with high prevalence of iron deficiency and anaemia. As anaemia is associated with extensive health effects, such as stunting, fatigue and impaired neurodevelopment reducing anaemia in infants is an urgent need in a global perspective. In a recently published observational study from Peru, anaemia at eight months of age was evaluated at infants born before and after a hospital change of regime from early to delayed cord clamping. The study resulted in a significant reduction of anaemia by 16% (from 75 to 59%) as well as a significant higher level of haemoglobin.

Rationale for Study in Nepal:

In Nepal, children age 6-17 months have high anaemia prevalence (72-78%). Approximately 50% of all anaemia among preschoolers can be contributed to ID. By performing the planned study in a country with high anaemia prevalence, we can reduce sample size dramatically and still be able to detect significant effects on haemoglobin levels and neurodevelopment.

Study Objective:

To evaluate the effects of delayed and early cord clamping on

1. Anaemia (and haemoglobin level) at 8 and 12 months
2. Ferritin at 8 and 12 months
3. Bilirubin at 2-3 days
4. Admission to the neonatal intensive care unit (NICU) or special care nursery
5. Development at 12 and 18-24 months of age.

Primary outcome:

The primary outcome will be infant haemoglobin 8 and 12 months of age.

Secondary outcomes:

The secondary outcome will be neonatal morbidity (need for phototherapy, and respiratory symptoms). Maternal postpartum haemorrhage; effects of delayed and early cord clamping on iron status at 8 and 12 months of age; psychomotor development at 12 months of age assessed by the Ages and Stages Questionnaire and development evaluated by The Bayley Scales of Infant and Toddler Development at 18-24 months.

Methods

Trial design and Participants:

Randomized controlled trial comparing delayed and early cord clamping will be implemented in the hospital. The study will be conducted at the Paropakar Maternity and Women's Hospital, Nepal.

Pregnant women are eligible if they meet the following criteria:

* Late preterm or term pregnancy (gestational age 34 to 41 weeks)
* Single pregnancy with expected vaginal delivery
* Mother/family give consent to return for follow-up at 8 and 12 months

Exclusion criteria are serious congenital malformations, syndromes, or other congenital diseases that could affect the outcome measures.

Intervention:

When delivery is imminent (expected within 10 minutes), the midwife will opened a sealed, numbered, opaque envelope containing the treatment allocation. The interventions consist of delayed clamping of the umbilical cord (≥180 seconds after delivery) or early clamping of the umbilical cord (≤60 s). The time from complete delivery of the baby to the first clamp on the umbilical cord will be measured with a stopwatch by the midwife's assistant or the surveillance officer. All other aspects of obstetric care will be managed according to standard practice at the hospital. In both groups, oxytocin will be given to the mother after the umbilical cord is clamped. All staff in the delivery unit will be trained in the study procedures before the trial started.

Follow-up:

After the delivery, the babies will be cared for according to clinical routines, and early breast feeding will be encouraged. As part of the study, the infant will be assessed at 1 and 6 hours by the midwife, who will record if the baby has been breast fed and the presence of respiratory symptoms (that is, respiratory rate >60 breaths/minute, presence of nostril flaring, grunting, or intercostal retractions).

Infants will stay at the postnatal ward with their mothers for two or three days, except for well babies whose mothers preferred to leave the hospital earlier and infants who requires admission to the neonatal unit. Transcutaneous bilirubin will be checked at 24 and 48 hours of age if newborn is still at the hospital, and before discharge.

At 8 and 12 months of age, infants will be scheduled for a follow-up visit including blood sampling (hemoglobin and ferritin) and weight and length measurements. Venous blood sampling will be performed. Before the visit, parents will be asked to complete a three day food diary to assess whether the infant was exclusively or partially breast fed and whether formula or solids were given. Parent will be assisted in answering the Ages & Stages Questionnaire.

If funding is achieved, children wil be examined by The Bayley Scales of Infant and Toddler Development, Third Edition at 18-24 months of age.

Physicians performing neonatal examinations, staff members responsible for collection of blood samples and background data, and laboratory staff performing analyses of blood samples will be blinded to each infant's allocation group.

Additional data collection:

The following information will be collected from maternal healthcare records: reported illness, medication, parity, weight, height, smoking habits at the time of admission.

Sample size:

The sample size for the primary outcome at eight months was estimated to find a difference of 15% (70% versus 55%) in the prevalence of anaemia between the two randomization groups with a power of 80% and a type I error rate of .05. Using Fisher's exact-test to analyze outcome data a group size of 176 would be needed. Taking into account an attrition rate of 35% we calculate to include 270 newborns in each group, i.e. a total of 540.

Ethical considerations:

All research involving newborn infants and small children need careful ethical considerations, mainly since the subjects themselves can't agree to whether they want to participate in the study or not. In particular, research that is not immediately of benefit for the patients needs ethical consideration. The included infants are healthy full-term infants undergoing umbilical cord clamping, which is a standard procedure after birth. The possible benefit of the intervention (delayed cord clamping) of increasing iron stores and preventing infant anaemia is estimated to be higher than the risk of probable adverse effects, such as hyperbilirubinaemia. Ethical approval has be sought and obtained from Nepal Health Research Council (June 6, 2014, 76/2014). Written informed parental consent will be obtained before the intervention, and parents can withdraw from the study at any time without any need for explanations.

Discussion and Policy Implication:

Reducing ID among infants is important as it is associated with impaired neurodevelopment. In Sweden, ID has been found among 26% of 12 months old infants. With high global prevalence of infant anaemia, delayed cord clamping has the potential to reduce infant anaemia and thereby improve infants' and children's health and development. In crude numbers, a reduction by 10% would mean an annual reduction of 60 000 infants with anaemia in Nepal. The trial is important to perform as although strong indications exists on the effect of delayed cord clamping on anaemia at 8 to 12 months of age, it has not been evaluated by a randomized trial. By the proposed study, outcome as well as safety effects will be analyzed, and results might not only contribute to the practice in Nepal, but also to the global community, in particular low income countries with a high prevalence of ID anaemia.

ELIGIBILITY:
Inclusion Criteria:

* Late preterm or term pregnancy (gestational age 34 to 41 weeks)
* Vaginal delivery

Exclusion Criteria:

* Serious congenital malformation, syndrome or other congenital disease that can affect the outcome measures

Ages: 34 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 540 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-12-11 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | 8 months plus/minus one month
  Hemoglobin will be analyzed be comparing means and as a categorical variable, defining anemia as Hemoglobin < 110 g/L

SECONDARY OUTCOMES:
Hemoglobin | 12 months plus/minus one month
  Hemoglobin will be analyzed be comparing means and as a categorical variable, defining anemia as Hemoglobin < 110 g/L
Ferritin | 8 months plus/minus one month
  Ferritin will be analyzed be comparing means and as a categorical variable, defining iron deficiency as Ferritin < 12 μg/L
Ferritin | 12 months plus/minus one month
  Ferritin will be analyzed be comparing means and as a categorical variable, defining iron deficiency as Ferritin < 12 μg/L
Iron deficiency anemia | 8 months plus/minus one month
  Defining iron deficiency as a combination of Hemoglobin < 110 g/L and Ferritin < 12 μg/L
Iron deficiency anemia | 12 months plus/minus one month
  Defining iron deficiency as a combination of Hemoglobin < 110 g/L and Ferritin < 12 μg/L
Bilirubin | 2 days
  Measured by a transcutaneous method.
Psychomotor development assessed by the Ages and Stages Questionnaire. | 12 months
  Ages and Stages Questionnaire is a parent report questionnaire available for developmental screening of children from one month to 5 ½ years. 30 questions are divided into 5 developmental domains (communication, gross motor, fine motor, problem solving and personal-social). Total score and scores within separate domains from the 48-month questionnaire will be assessed.
Psychomotor development assessed by Bayley Scales of Infant and Toddler Development 3rd ed. (Bayley III) | 18 months plus 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ola Andersson, MD PhD, Principal Investigator — Uppsala University; Ashish KC, MD, Principal Investigator — Uppsala University
Locations (1):
- Paropakar Maternity and Women's Hospital, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson O, Hellstrom-Westas L, Andersson D, Domellof M. Effect of delayed versus early umbilical cord clamping on neonatal outcomes and iron status at 4 months: a randomised controlled trial. BMJ. 2011 Nov 15;343:d7157. doi: 10.1136/bmj.d7157. PMID 22089242
- [Background] Andersson O, Domellof M, Andersson D, Hellstrom-Westas L. Effect of delayed vs early umbilical cord clamping on iron status and neurodevelopment at age 12 months: a randomized clinical trial. JAMA Pediatr. 2014 Jun;168(6):547-54. doi: 10.1001/jamapediatrics.2013.4639. PMID 24756128
- [Result] Kc A, Rana N, Malqvist M, Jarawka Ranneberg L, Subedi K, Andersson O. Effects of Delayed Umbilical Cord Clamping vs Early Clamping on Anemia in Infants at 8 and 12 Months: A Randomized Clinical Trial. JAMA Pediatr. 2017 Mar 1;171(3):264-270. doi: 10.1001/jamapediatrics.2016.3971. PMID 28114607
- [Result] Rana N, Kc A, Malqvist M, Subedi K, Andersson O. Effect of Delayed Cord Clamping of Term Babies on Neurodevelopment at 12 Months: A Randomized Controlled Trial. Neonatology. 2019;115(1):36-42. doi: 10.1159/000491994. Epub 2018 Oct 2. PMID 30278462
- [Result] Rana N, Ranneberg LJ, Malqvist M, Kc A, Andersson O. Delayed cord clamping was not associated with an increased risk of hyperbilirubinaemia on the day of birth or jaundice in the first 4 weeks. Acta Paediatr. 2020 Jan;109(1):71-77. doi: 10.1111/apa.14913. Epub 2019 Jul 15. PMID 31240753
- [Derived] Berg JHM, Isacson M, Basnet O, Gurung R, Subedi K, Kc A, Andersson O. Effect of Delayed Cord Clamping on Neurodevelopment at 3 Years: A Randomized Controlled Trial. Neonatology. 2021;118(3):282-288. doi: 10.1159/000515838. Epub 2021 May 7. PMID 33965945
- [Derived] Kc A, Malqvist M, Rana N, Ranneberg LJ, Andersson O. Effect of timing of umbilical cord clamping on anaemia at 8 and 12 months and later neurodevelopment in late pre-term and term infants; a facility-based, randomized-controlled trial in Nepal. BMC Pediatr. 2016 Mar 10;16:35. doi: 10.1186/s12887-016-0576-z. PMID 26965317